CLINICAL TRIAL: NCT03430310
Title: Return of First-phase Insulin Secretion in Type 2 Diabetes is Associated With Depletion of Pancreas Lipid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Barbara Gower, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DK116726 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-02-12 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycemic Diet (Experimental): The investigators will use a Low Glycemic Load Diet (LG Diet), which emphasizes low-glycemic sources of carbohydrate, and includes mainly whole foods (vegetables, fruits, whole grains) with minimal highly processed grain products and added sugar. Protein foods will include meat, poultry, fish, eggs, and whey protein supplements if necessary (e.g., for vegetarians). Fat-containing foods will include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; avocados; and the fat found in meat. A number of full-fat dairy products will be included. Saturated fat from red meat will be limited to less than 10% of daily caloric intake. Participants will obtain the majority of their fat intake from mono-unsaturated fatty acids (e.g. olive oil), and medium-chain triglycerides (e.g., coconut oil and cream); from nuts and nut butters; and from fresh fish.
  Interventions: Other: Low Glycemic Diet
- Control Diet (Placebo Comparator): The Control diet will be compatible with both the American Diabetes Association and The United States Department of Agriculture guidelines. Participants will be given low-fat foods, whole-grain foods, fruits, and vegetables. The meal plans will minimize cholesterol, high-fat foods, high-cholesterol foods, processed starches, and added sugar, and will provide <2300 mg/day sodium. Saturated fat will be limited to less than 10% of total energy, and all dairy products will be fat-free (or low-fat). Although the Control diet will be a healthful diet, it will include a greater amount of carbohydrate foods from such sources as bread, potatoes, and pasta that will distinguish it qualitatively from the LG diet. In addition, it will have quantitatively more total energy from carbohydrate than the LG diet.
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: Low Glycemic Diet — The investigators will use a Low Glycemic Load Diet (LG Diet), which emphasizes low-glycemic sources of carbohydrate, and includes mainly whole foods (vegetables, fruits, whole grains) with minimal highly processed grain products and added sugar. Protein foods will include meat, poultry, fish, eggs, and whey protein supplements if necessary (e.g., for vegetarians). Fat-containing foods will include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; avocados; and the fat found in meat. A number of full-fat dairy products will be included. Saturated fat from red meat will be limited to less than 10% of daily caloric intake. The participants will obtain the majority of their fat intake from mono-unsaturated fatty acids (e.g. olive oil), and medium-chain triglycerides (e.g., coconut oil and cream); from nuts and nut butters; and from fresh fish.
  Arms: Low Glycemic Diet
Other: Control Diet — The Control diet will be compatible with both the American Diabetes Association and The United States Department of Agriculture guidelines. Participants will be given low-fat foods, whole-grain foods, fruits, and vegetables. The meal plans will minimize cholesterol, high-fat foods, high-cholesterol foods, processed starches, and added sugar, and will provide <2300 mg/day sodium. Saturated fat will be limited to less than 10% of total energy, and all dairy products will be fat-free (or low-fat). Although the Control diet will be a healthful diet, it will include a greater amount of carbohydrate foods from such sources as bread, potatoes, and pasta that will distinguish it qualitatively from the LG diet. In addition, it will have quantitatively more total energy from carbohydrate than the LG diet.
  Arms: Control Diet

SUMMARY:
The hypothesis for this study is that pancreas lipid will be more closely associated with first-phase beta-cell response in African-Americans than in European-Americans, both at baseline and in response to treatment. The investigators will determine whether race influences the association of pancreas lipid with beta-cell function.The proposed research builds upon the investigators preliminary observations in non-diabetic adults that reduction in dietary glycemic load, in the absence of weight loss, selectively reduces visceral adipose tissue and ectopic lipid, and is associated with improvements in insulin sensitivity and beta-cell function. No study has attempted to test the hypothesis that selective reduction in pancreatic lipid with a simple change in diet composition, in the absence of energy restriction, will lead to the recovery of beta-cell function in patients with early Type 2 Diabetes (T2D). The investigators hypothesize that participants following a Low Glycemic Diet will show a greater decrease in pancreas lipid. Specifically, the investigators will be the first to demonstrate that a weight-maintaining low-glycemic diet improves glucose tolerance by increasing first-phase insulin secretion. Results may be particularly relevant to African-Americans who are at greater risk for T2D.

DETAILED DESCRIPTION:
The decline in first-phase insulin secretion is a key event in the etiology of type 2 diabetes (T2D). Although the cause of beta-cell failure is not clear, "lipotoxicity" has been proposed. Bariatric surgery and very-low calorie diets in patients with T2D induce disease remission, characterized by a return of first-phase insulin secretion and a depletion of pancreas lipid. However, these are extreme approaches to treating T2D, and non-invasive, sustainable, yet equally effective, treatments are needed. The investigators have shown in individuals at risk for T2D that an intervention with a weight-maintaining low-glycemic (LG) diet selectively depletes visceral adipose tissue and ectopic lipid in muscle while preserving thigh subcutaneous adipose and lean body mass. This observation suggests that such diets are able to "remodel" body composition by re-partitioning energy away from metabolically harmful lipid stores. Participants on the LG diet also demonstrated improved insulin sensitivity and a dramatic (9-fold) increase in first-phase insulin secretion. Thus, the investigators hypothesize that a weight-maintaining LG diet will selectively deplete ectopic adipose tissue, including pancreatic lipid, and will permit recovery of beta-cell function in individuals with T2D. Rescue of beta-cell function may be particularly important in African-Americans (AA), who as a group demonstrate a high prevalence of T2D, for reasons that cannot be explained by lifestyle. AA are likely to be vulnerable to beta-cell failure due to inherently high beta-cell responsiveness (demonstrable in healthy young children). Further, it has been shown that pancreas lipid is a determinant of prediabetes specifically in AA. Thus, the investigators hypothesize that an LG diet will be particularly beneficial to beta-cell function and glycemic control among AA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes within the past 10 years
* Treated with diet, Metformin, or dipeptidyl peptidase 4 (DPP-IV) inhibitors
* Adult men and women age 35-65 yr
* Have a Hemoglobin A1c <7.0
* African American or European American race
* Will be overweight (BMI 25-45 kg/m2) but have a stable BMI (<5 kg change in the past 6 months)

Exclusion Criteria:

* Use of glucocorticoids
* Estimated glomerular filtration rate <60
* Alanine aminotransferase >2.5-fold above the normal upper limit
* Tobacco or recreational drug use
* Unable to undergo MRI

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was between September 2018 and March 2023. Recruitment methods included flyers, local advertisements, radio, tv, social media, and word of mouth.
Pre-assignment Details: No washout or run-in was used for this study.
Groups:
- Low Glycemic Diet: The investigators will use a Low Glycemic Load Diet (LG Diet), which emphasizes low-glycemic sources of carbohydrate. Protein foods will include meat, poultry, fish, eggs, and whey protein supplements if necessary (e.g., for vegetarians). Fat-containing foods will include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; avocados; and the fat found in meat. A number of full-fat dairy products will be included. Saturated fat from red meat will be limited to less than 10% of daily caloric intake. Participants will obtain the majority of their fat intake from mono-unsaturated fatty acids (e.g. olive oil), and medium-chain triglycerides (e.g., coconut oil and cream); from nuts and nut butters; and from fresh fish.
Period: Overall Study
Arm/Group | Low Glycemic Diet | Control Diet
Started | 32 | 33
Completed | 27 | 30
Not Completed | 5 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — COVID shutdown March 2020 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Glycemic Diet | Control Diet | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 31 | 63
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 6 | 8 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 12 | 11 | 23
  African American | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.94 (6.06) | 35.90 (6.60) | 35.43 (6.31)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Liver Fat
Description: Assessing the overall percentage of liver fat with magnetic resonance imaging (MRI) to measure
Time Frame: Baseline, week 12
Measure: Mean (Standard Error); unit: percent liver fat
Arm/Group | Low Glycemic Diet | Control Diet
Number analyzed (Participants) | 27 | 30
percent liver fat | 5.4 (0.7) | 7.3 (0.6)
Statistical Analysis 1: Comparison: Low Glycemic Diet vs Control Diet; Test type: Superiority; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Low Glycemic Diet | Control Diet
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

LIMITATIONS AND CAVEATS:
Repository information has been uploaded into document section as requested by JCEM.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT03430310/Prot_SAP_000.pdf